CLINICAL TRIAL: NCT03325179
Title: A Clinical Trial of Acupoint Thread-embedding Therapy for Simple Obesity
Brief Title: A Clinical Trial of Thread-embedding Therapy at Acupuncture Point for Simple Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: shutcmidd
Record Dates: First submitted 2017-09-03; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-06

CONDITIONS: Weight Loss; Simple Obesity
Keywords: Simple Obesity; Thread-embedding Therapy; Acupuncture
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants received treatment (Experimental): 100 participants who are diagnosed as simple obesity under the standards of... are planned to enrolled in the trial. Each will receive Thread-embedding therapy.
  Interventions: Other: Thread-embedding Therapy

INTERVENTIONS:
Other: Thread-embedding Therapy

SUMMARY:
Thread-embedding Therapy has been used for treating Obesity in recent years. This research is aimed to observe the clinical effect of thread-embedding therapy in treating Simple Obesity. One hundred patients is planned to be enrolled in the research and receive a thread-embedding therapy. The level of BMI, serum triglyceride, cholesterol and fasting blood glucose will be adopted for evaluation before and after therapy.

DETAILED DESCRIPTION:
Each participant will receive thread-embedding therapy every two weeks, and eight times in all.Blood test will be taken at the beginning of the first week of the whole therapy, and at the end of the 8th therapy. During the periods of whole therapy, the participants shall follow diets control and physical exercise as the protocol described.

ELIGIBILITY:
Inclusion Criteria:

* patients with age from 18 to 60 years old;
* patients with BMI≥ 24, meanwhile waist more than 85 cm (for male) or 80 cm (for female);
* patients with diagnosed as central adiposity and/or Simple obesity according to the diagnosis criteria；
* patients who is willing to cooperate with the test treatment and signed informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* patients who Syncope after acupuncture；
* patients who present hypersensitivity reactions after acupoint-embedding therapy;
* patients with serious heart, liver, kidney, brain and other diseases;
* patients with severe primary diseases;
* patients with psychiatric diseases；
* patients who did not meet the criteria for the inclusion criteria while investigators find out during the trial;
* participants who did not complete dietary control and physical exercise as the protocol described.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
The change Body Weight | participants will receive Thread-embedding Therapy twice a week lasting for 16 weeks subsequently.8 times in all.
  a 5 percent of loss of body weight will be judged as effective

SECONDARY OUTCOMES:
The effection on cholesterol | Therapy is the same as mentioned above. Participants will take blood test at the beginning of the first week of the therapy, and at the end of the 16th week.
  a target examined by blood test, in order to compare the Lipid metabolism
The effection on triglyceride | Therapy is the same as mentioned above. Participants will take blood test at the beginning of the first week of the therapy, and at the end of the 16th week.
  a target examined by blood test, in order to compare the Lipid metabolism
The effection on fasting blood glucose | Therapy is the same as mentioned above. Participants will take blood test at the beginning of the first week of the therapy, and at the end of the 16th week.
  to compare the level of glucose in order to get the message of improvement of blood glucose disorder by our therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Digestive Diseases of Longhua Hospital affiliate to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China